CLINICAL TRIAL: NCT01260623
Title: In Vivo Prednisolone/Prednisone Pharmacokinetic Pilot Study in Children With Asthma Exacerbations
Brief Title: Pilot Study of How Children With Asthma Exacerbations Metabolize Prednisone
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: R-09-406; 16380 (Other: REB)
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Asthma Exacerbation
Keywords: asthma; pharmacokinetics; prednisone; prednisolone; asthma exacerbation; pharmacokinetic profile
MeSH Terms: conditions — Asthma | interventions — Prednisolone; Prednisone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prednisolone and prednisone — oral, or intravenous prednisone, prednisolone, given the first time for asthma exacerbation

SUMMARY:
The objective of the investigators pilot study is to assess the pharmacokinetic profile of two corticosteroid drugs, prednisone and prednisolone, in children who present to the pediatric emergency department with an asthma exacerbation. The investigators hypothesis is that the pharmacokinetic profile in this population will be similar to healthy children and adults.

DETAILED DESCRIPTION:
The standard of practice in treating children with asthma exacerbations is to give corticosteroid drugs early in the course of the exacerbation. These drugs decrease symptoms, provide faster time to recovery and improve of quality of life. However, there is 100% variability in a child's response to corticosteroids at a standard dose which is based on primarily on adult studies. The pharmacokinetic analysis or the process by which a drug is metabolized by the body is the first step to determine the proper dose.

Patients between the ages of 2 and 16 years with asthma exacerbations will be recruited from the pediatric emergency department. After the patients get the drugs, blood samples will be drawn over 8 hours to get the following parameters: maximum concentration reached in the body, the time for the drug to be eliminated from the body, how long the drug stays in the body, how much of the drug is found in the urine after it is given, and concentration of metabolites or breakdown products in urine and blood. These are the parameters needed to make the pharmacokinetic profile and is the first step towards appropriate dosing of these two medications for asthma exacerbations in children.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 2 to 16 years
* acute asthma exacerbation requiring an oral corticosteroid (either prednisone or prednisolone)
* any "reactive airways disease" treated like asthma

[Asthma is defined as at least 2 wheezing episodes and/or the patient has been treated with beta agonist and/or inhaled, oral or intravenous corticosteroids for the recurrent episodes of wheezing in the past] [Acute asthma exacerbation is defined as wheezing episode with any of the following symptoms: tachypnea, dyspnea, use of accessory muscles, or an increased need for short acting beta agonist prior to presentation to PED]

Exclusion Criteria:

* any systemic corticosteroid use within 1 week of presentation to PED
* use of any other corticosteroid apart from oral prednisone or prednisolone for the current acute asthma exacerbation
* bronchiolitis
* underlying chronic medical condition other than asthma (ie: cystic fibrosis, nephrotic syndrome, epilepsy, etc)
* liver impairment (including elevated transaminases)
* renal impairment
* primary or secondary immunodeficiences
* concomitant immunosuppressive medication use
* IVIG use within 4 weeks
* need for assisted ventilation

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children between the ages of 2 and 16 years who present to the tertiary care pediatric emergency department in London, Ontario with an asthma exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-09-09 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic profile of prednisone and prednisolone | over 8 hours post ingestion of medication
  The children will receive prednisone or prednisolone by mouth at current standard dose of 1mg/kg. Blood samples will be drawn from the catheter at baseline (0 hours), 1, 2, 4, 6, and 8 hours post ingestion of the medication. All samples will be analyzed for prednisone and prednisolone concentrations, and breakdown product concentrations. Urine samples will be collected prior to discharge for analysis of fractional excretion of prednisone, prednisolone, and the metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rieder, MD, Ph.D, FRCPC, Principal Investigator — Pediatric Emergency Dept, Children's Hospital, London Health Sciences Centre
Locations (1):
- Pediatric Emergency Department, Children's Hospital, London Health Sciences Centre, London, Ontario, Canada